CLINICAL TRIAL: NCT04620434
Title: Improvement of the Glottic View by the Use of Video Laryngoscope
Brief Title: Improvement of the Glottic View by Video Laryngoscope
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Dongwook Won, Associate professor, Seoul National University Hospital
Other Study IDs: 30-2020-25
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Laryngoscope; Intubation; Laryngoscopy
Keywords: Video laryngoscope; Glottis; Airway

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient: 39 patients who are planning surgeries that require general anesthesia and tracheal intubation
  Interventions: Device: Video laryngoscopic view; Device: Direct laryngoscopic view

INTERVENTIONS:
Device: Video laryngoscopic view — The glottic view on the screen of the video laryngoscope during laryngoscopy with a C-MAC video laryngoscope, which installed with Macintosh blade.
Device: Direct laryngoscopic view — The glottic view evaluated by the anesthesiologist who performing tracheal intubation, by direct laryngoscopy with C-MAC installed with Macintosh blade.

SUMMARY:
This study aims to compare the exposure of glottis by the use of video and direct laryngoscopy.

DETAILED DESCRIPTION:
It is well known that a video laryngoscope can provide better glottic view than a direct laryngoscope. However, to date, a direct laryngoscope has been the standard equipment for tracheal intubation. Recently, it seems that use of the video laryngoscope has increased. However, the advantage of the video laryngoscope over a direct laryngoscope has not been measured quantitatively. In this study, the glottic view by the use of video laryngoscope will be compared with that of the direct laryngoscope simultaneously, by using C-MAC S-imager installed with a disposable Macintosh blade. Intubating anesthesiologists will use it as if it is a direct laryngoscope. Simultaneously, the glottic views visualized on the monitor of the video laryngoscope will be recorded and evaluated later. For quantitative comparison, the glottic view will be scored with the Percentage of glottic opening scale, for both direct laryngoscopy and video laryngoscopy. Also, the glottic view will be compared by Cormack-Lehane grade.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are over 18 years old, and are planning surgeries that require general anesthesia and tracheal intubation.

Exclusion Criteria:

* Patients who are not agreed to participate in the trial
* Patients who have a poor dental condition which requires other than direct laryngoscopy
* Patients who require rapid sequence induction technique
* Patients with cervical spine instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have airways with various degrees of difficulty will be candidates for this observational study.
Sampling Method: Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
POGO (Percentage of Glottic Opening) score | during laryngoscopy
  POGO (Percentage of Glottic Opening) score of the glottic view by video/direct laryngoscope during laryngoscopy without external laryngeal manipulation. (Percentage of glottic opening score, which means a better outcome at higher score: linear span from the anterior commissure to the interarytenoid notch; 0%, only interarytenoid notch seen; 100% full view of vocal cords)
Cormack-Lehane grade | during laryngoscopy
  Cormack-Lehane grade with video/direct laryngoscope, during laryngoscopy without external laryngeal manipulation (Cormack-Lehane grade, which means a better outcome at lower score: grade 1, Full view of glottis; grade 2a, Partial view of glottis; grade 2b, Only posterior extremity of glottis or arytenoid cartilages; grade 3, Only epiglottis seen; grade 4, Neither glottis nor epiglottis seen)

SECONDARY OUTCOMES:
POGO score with external laryngeal manipulation | during laryngoscopy
  POGO score of the glottic view by video/direct laryngoscope during laryngoscopy with external laryngeal manipulation. (Percentage of glottic opening score, which means a better outcome at higher score: linear span from the anterior commissure to the interarytenoid notch; 0%, only interarytenoid notch seen; 100% full view of vocal cords)
Cormack-Lehane grade with external laryngeal manipulation | during laryngoscopy
  Cormack-Lehane grade with video/direct laryngoscope, during laryngoscopy with external laryngeal manipulation. (Cormack-Lehane grade, which means a better outcome at lower score: grade 1, Full view of glottis; grade 2a, Partial view of glottis; grade 2b, Only posterior extremity of glottis or arytenoid cartilages; grade 3, Only epiglottis seen; grade 4, Neither glottis nor epiglottis seen)

CONTACTS AND LOCATIONS:
Overall Officials: Dongwook Won, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- SMG-SNU, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arulkumaran N, Lowe J, Ions R, Mendoza M, Bennett V, Dunser MW. Videolaryngoscopy versus direct laryngoscopy for emergency orotracheal intubation outside the operating room: a systematic review and meta-analysis. Br J Anaesth. 2018 Apr;120(4):712-724. doi: 10.1016/j.bja.2017.12.041. Epub 2018 Feb 26. PMID 29576112
- [Background] Kaplan MB, Hagberg CA, Ward DS, Brambrink A, Chhibber AK, Heidegger T, Lozada L, Ovassapian A, Parsons D, Ramsay J, Wilhelm W, Zwissler B, Gerig HJ, Hofstetter C, Karan S, Kreisler N, Pousman RM, Thierbach A, Wrobel M, Berci G. Comparison of direct and video-assisted views of the larynx during routine intubation. J Clin Anesth. 2006 Aug;18(5):357-62. doi: 10.1016/j.jclinane.2006.01.002. PMID 16905081
- [Background] Levitan RM, Ochroch EA, Kush S, Shofer FS, Hollander JE. Assessment of airway visualization: validation of the percentage of glottic opening (POGO) scale. Acad Emerg Med. 1998 Sep;5(9):919-23. doi: 10.1111/j.1553-2712.1998.tb02823.x. PMID 9754506
- [Background] Cormack RS, Lehane J. Difficult tracheal intubation in obstetrics. Anaesthesia. 1984 Nov;39(11):1105-11. PMID 6507827